CLINICAL TRIAL: NCT02761486
Title: Pilot Trial to Examine the Effect of Aspirin on the Gut Microbiome
Brief Title: Effect of Aspirin on Gut Microbiome
Acronym: ASMIC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2016NTLS049; 2016NTLS049 (Other: UMN Clinical Protocol Review Committee)
Record Dates: First submitted 2016-04-29; First posted 2016-05-04 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: aspirin; gut microbiome; inflammation; placebo; circulating biomarker
MeSH Terms: conditions — Inflammation | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aspirin (Active Comparator): The subjects will receive 325 mg of aspirin once a day for 6 weeks followed by a 6-week washout.
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): The subjects will receive placebo once a day for 6 weeks followed by a 6-week washout.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — 325mg aspirin per day
  Other Names: Acetylsalicylic acid (ASA)
  Arms: Aspirin
Drug: Placebo — placebo in matching capsules
  Arms: Placebo

SUMMARY:
Regular use of aspirin may reduce the incidence of colorectal cancer (CRC). However, it is unclear through which mechanism aspirin exerts its effect, in whom it decreases CRC risk and in whom it causes side effects. Recently, the imbalanced gut microbiome was linked to inflammation and CRC risk. The main hypothesis for this study is that aspirin may decrease CRC risk via targeting the gut microbiome. The study will be a randomized placebo-controlled double-blinded design, recruiting 50 healthy subjects, 50-75 years old, from the PRospective Evaluation of SEPTin 9 (PRESEPT) cohort living in the greater Twin Cities area, who will receive either aspirin or placebo for 6 weeks.

DETAILED DESCRIPTION:
The pilot study will evaluate the feasibility of conducting a large randomized trial and estimate the effects of aspirin on the gut microbiome. The study will recruit 50 healthy subjects, 50-75 years old, from the PRospective Evaluation of SEPTin 9 (PRESEPT) cohort living in the greater Twin Cities area.

The Primary Aim is to estimate the impact of a 3- and 6-week intake of once daily 325 mg aspirin on the composition of the gut microbiome using a randomized placebo-controlled double-blinded design, i.e. examine the change of microbiome over time within and between the subjects. The hypothesis for this aim is that in the aspirin arm versus the placebo arm, gut microbiome composition will shift towards a lower proportion of pro-inflammatory, CRC-predisposing bacteria (e.g. Fusobacteria) and higher proportion of anti-inflammatory, CRC-protective bacteria (e.g. butyrate-producing bacteria).

The Secondary Aims are to examine the correlation between the aspirin-related changes in microbiome profile with the levels of circulating inflammatory biomarkers in urine and plasma. Within-individual and between-arm differences in microbiome composition will be compared after 3 and 6 weeks of aspirin intake. Also, the microbiome composition will be compared after 3-week and 6-week wash-out periods to test whether these periods are sufficient to restore gut microbiome composition to a pre-treatment level. This study will inform future crossover randomized studies focusing on CRC preventive interventions that will enable clinicians to identify optimal candidates for aspirin therapy for the purposes of CRC prevention using this accessible and cheap drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 50-75 years who reside within the greater Twin Cities area
* Capable and willing to comply with the entire study protocol
* Able to give voluntary written informed consent.

Exclusion Criteria:

* Use of any aspirin-containing products or other non-steroidal anti-inflammatory drugs (NSAIDs) (≥ 2 days per week on a regular basis)
* Known hypersensitivity to NSAIDs
* Any active cancer, history of gastrointestinal cancer, or chronic disease such as peptic ulcer, irritable bowel syndrome, inflammatory bowel disease, intestinal malabsorption syndrome or other gastrointestinal disorder
* History of any coagulation, bleeding, or blood disorders (e.g. Anemia)
* History of stroke/ Transient Ischemic Attack
* Acute heart disease or history of heart attack, atrial fibrillation, or angina
* Diagnosis of dementia
* Use of antibiotics, antiplatelets (e.g. clopidogrel), or anticoagulants (e.g. warfarin) within the last 3 months. A complete list of contraindicated medications will be provided (Appendix A)
* Regular use of laxatives (e.g. Ex-lax, Dulcolax, Miralax) that may affect the microbiome ≥2 days a week (Appendix B)
* Body mass index (BMI) greater than or equal to 40 or less than or equal to 17 kg/m2 at screening visit
* Unexplained change in weight (>4.5 kg) within the past 6 months
* Major changes in eating habits within the past 3 months

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Composition of the gut microbiome | 5 times within 12 weeks
  Fecal microbial diversity and the prevalence of specific taxa associated with colorectal cancer (e.g. Fusobacteria, butyrate producing bacteria) will be estimated at each time point. The aspirin-related changes in the prevalence of each taxon will be assessed individually and also combined into a microbiome index (the abundance of protective taxa will be included as a negative value).

SECONDARY OUTCOMES:
Urinary and blood inflammatory biomarkers | 2 times within 6 weeks
  Each inflammatory biomarker (e.g. urinary metabolite of Prostaglandin E2 (PGE2)) will be measured before and after treatment with aspirin. Changes in inflammatory markers will be correlated to changes in the microbial diversity and the microbiome index.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Prizment, PhD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- Epidemiology Clinical Research Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No. The results of the study will be disseminated to various stakeholders through the publication of a manuscript in a peer-reviewed journal and through presentation at scientific meetings.